CLINICAL TRIAL: NCT04138992
Title: a Prospective Random Study on the Efficacy and Safety of Bevacizumab in Untreated Patients With Locally Advanced Cervical Cancer
Brief Title: A Study on the Efficacy and Safety of Bevacizumab in Untreated Patients With Locally Advanced Cervical Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Mei Shi, head of department, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJFL-2019-01-LACC-bevacizumab
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Disease Free Survival
Keywords: Bevacizumab; local advanced cervical cancer; concurrent chemoradiotherapy
MeSH Terms: interventions — Bevacizumab; Cisplatin; Docetaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- study group A (Experimental): bevacizumab combined with neoadjuvant chemotherapy and concurrent chemoradiotherapy：
  1. bevacizumab combined with neoadjuvant chemotherapy for 2 cycles: Bevacizumab will be used as 7.5 mg/kg, once every three weeks; DDP 75mg/m2, intravenous injection，once three week; Docetaxel 75mg/m2, intravenous injection，once three week;
  2. bevacizumab combined with concurrent chemoradiotherapy: Bevacizumab will be used as 7.5 mg/kg, once every three weeks; DDP 75mg/m2, intravenous injection，once three week pelvic radiotherapy will be delivered with 45-50Gy/25f; enlarged lymph nodes be irradiated by 62.5Gy/25f with sib-IMRT; brachytherapy be delivered to cervix and primary tumor
  Interventions: Drug: bevacizumab; Drug: DDP; Drug: Docetaxel; Radiation: radiotherapy
- study group B (Experimental): study arm: bevacizumab combined with concurrent chemoradiotherapy： Bevacizumab will be used as 7.5 mg/kg, once every three weeks; DDP 75mg/m2, intravenous injection，once three week; pelvic radiotherapy will be delivered with 45-50Gy/25f; enlarged lymph nodes be irradiated by 62.5Gy/25f with sib-IMRT; brachytherapy be delivered to cervix and primary tumor
  Interventions: Drug: bevacizumab; Drug: DDP; Radiation: radiotherapy
- control (Active Comparator): standard concurrent chemoradiotherapy: DDP 40mg/m2, intravenous injection，once a week; pelvic radiotherapy will be delivered with 45-50Gy/25f; enlarged lymph nodes be irradiated by 62.5Gy/25f with sib-IMRT; brachytherapy be delivered to cervix and primary tumor
  Interventions: Drug: DDP; Radiation: radiotherapy

INTERVENTIONS:
Drug: bevacizumab — bevacizumab will be used during neoadjuvant and concurrent chemoradiotherapy
  Other Names: Avastin
  Arms: study group A; study group B
Drug: DDP — DDP will be used during neoadjuvant and concurrent chemoradiotherapy
  Other Names: Cisplatin
Drug: Docetaxel — used in neoadjuvant chemotherapy
  Arms: study group A
Radiation: radiotherapy — standard treatment includes pelvic external beam radiation and brachytherapy
  Other Names: RT

SUMMARY:
To verify the clinical efficacy and safety of bevacizumab in treating local advanced cervical cancer, present study was designed to investigate the clinical results of bevacizumab combined with concurrent chemoradiotherapy (CCRT) in local advanced cervical cancer

DETAILED DESCRIPTION:
Cervical cancer is the most common malignant tumor of the female productive system in developing countries and regions. Since five large-sample randomized controlled clinical trials have reported that concurrent chemoradiotherapy can improve the survival rate of patients with cervical cancer in the early 20th century, cisplatin-based concurrent chemoradiotherapy has become the standard treatment for locally advanced cervical cancer (LACC) . LACC has the characteristics of high invasiveness, high lymphatic metastasis and poor prognosis. The size and stage of the tumor are two independent prognostic factors. In 2008, a retrospective study published in Journal of Clinical Oncology(JCO) suggested that single-agent concurrent chemoradiotherapy did not improve disease-free survival (DFS) or overall survival (OS) for patients with FIGO stage II-IVA tumors. Multiple studies reported poor prognosis in patients with primary tumors whose diameters were larger than 4 cm, 5 cm or 6 cm , and in 2016, Fokdal. et al. reported a low local control rate if the residual tumor volume was larger than 30 cc prior to afterloading brachytherapy . In the EMBRACE trial, Jastaniyah et al. divided tumors into five groups based on the difference between the tumor volume before treatment and prior to afterloading brachytherapy, and found that the dose coverage of the HR-CTV by D90 was low for patients with a large primary tumor volume and a poor treatment response [13]. Therefore, for patients with a large primary tumor volume, further studies are required to investigate whether accelerated tumor volume regression prior to afterloading brachytherapy is meaningful to escalating the local afterloading dose delivered to tumor and improving the local control rate and OS.

In recent years, with the rapid development of molecular biology, there have been multiple clinical trials regarding the molecular targeted drug therapy for tumor cell-specific targets . The angiogenesis inhibitor, bevacizumab, is the first molecular targeted drug for recurrent or advanced cervical cancer, which inhibits tumor angiogenesis by blocking the function of the vascular endothelial growth factor (VEGF). In a GOG phase II clinical trial, bevacizumab was applied to 46 patients with recurrent cervical cancer. The study reported a progression-free survival (PFS) of more than 6 months, with a median PFS and a median OS of 3.50 months and 7.29 months, respectively. Another GOG240 phase III clinical trial showed that chemotherapy combined with bevacizumab extended the OS of patients with recurrent and metastatic cervical cancer. United States' NCCN Clinical Practice Guidelines recommend the combined use of bevacizumab with paclitaxel + cisplatin for the first-line treatment of current and metastatic cervical cancer. However, there is a lack of evidence for the use of bevacizumab in the treatment of LACC.

The above background information raises the questions of: during the initial treatment of LACC, can the introduction of bevacizumab improve the patient's tumor regression rate and OS? And compared to concurrent chemoradiotherapy directly combined with bevacizumab, can neoadjuvant chemotherapy combined with bevacizumab + concurrent chemoradiotherapy further improve the therapeutic outcome? However, currently there is no research on these topics. In 2017, our research team reported poor prognosis in patients with LACC who had a high VEGFR expression . This result indicated that anti-angiogenic therapy could benefit patients with LACC. To investigate the clinical efficacy and safety of bevacizumab in treating local advanced cervical cancer, we design this clinical study

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven, invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix
2. 2018FIGO clinical stage I-IIIC disease

Exclusion Criteria:

1， Prior invasive malignancy (except non-melanomatous skin cancer), unless disease free for a minimum of 3 years; 2， Prior systemic chemotherapy within the past three years; 3， Prior radiotherapy to the pelvis or abdomen ; 4， Distant metastasis; 5， Severe, active co-morbidity; 6， patients with FIGO stage IVA 7， Bevacizumab is prohibited to the patients with active bleeding and hypertension

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3 year
  disease free survival

SECONDARY OUTCOMES:
local control | 3 year
  local control

OTHER OUTCOMES:
distant metastasis | 3 year
  distant metastasis
grade 3-4 side effects | 3 year
  grade 3-4 side effects

CONTACTS AND LOCATIONS:
Overall Officials: mei shi, M.D., Principal Investigator — Xijing Hospital
Locations (1):
- Department of Radiation Oncology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- See also: Bevacizumab — http://ncbi.nlm.nih.gov